CLINICAL TRIAL: NCT00312650
Title: A Phase II Study of Every 2 Week Doxil and Gemcitabine in Recurrent Ovarian Cancer
Brief Title: Doxil and Gemcitabine in Recurrent Ovarian Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: Ortho Biotech, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-0120
Record Dates: First submitted 2006-04-06; First posted 2006-04-10 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Ovarian Carcinoma
Keywords: ovarian cancer; recurrent; progressive
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — liposomal doxorubicin; Gemcitabine

INTERVENTIONS:
Drug: liposomal doxorubicin and gemcitabine

SUMMARY:
Standard treatment for recurrent ovarian cancer is chemotherapy with one or more drugs. One of these drugs, Doxil, can cause skin toxicity at the standard dosages. This study investigates using a lower dose given more frequently in combination with a second drug Gemcitabine.

DETAILED DESCRIPTION:
This study will evaluate the toxicities of Doxil and Gemcitabine given on an every two week basis. Our hypothesis is that toxicity will be less than that with standard dosing without any negative effect on survival. Patients will also be evaluated with CT scans every 3 months. Toxicity will be assessed with every cycle of treatment. Treatment will continue until toxicity or signs of progression.

ELIGIBILITY:
Inclusion Criteria:

* recurrent platinum resistant ovarian cancer
* measurable disease

Exclusion Criteria:

* prior treatment with Doxil or Gemzar
* life expectancy <3months
* cardiac ejection fraction <50%

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2006-04; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
rate of hand-foot syndrome

SECONDARY OUTCOMES:
objective response rate

CONTACTS AND LOCATIONS:
Overall Officials: Paul A DiSilvestro, MD, Principal Investigator — Program in Women's Oncology
Locations (1):
- Women and Infants' Hospital, Providence, Rhode Island, United States